CLINICAL TRIAL: NCT02242097
Title: A Phase II Clinical Trial Evaluating Ibrutinib Maintenance Following Intensive Induction for Patients With Previously Untreated Mantle Cell Lymphoma (MCL)
Brief Title: Ibrutinib After Intensive Induction in Treating Patients With Previously Untreated Mantle Cell Lymphoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 14H06; NCI-2014-01777 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PCI-32765MCL2003; STU00098385; NU 14H06 (Other: Northwestern University); P30CA060553 (NIH)
Record Dates: First submitted 2014-09-12; First posted 2014-09-16 (Estimated); Results first posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-02

CONDITIONS: Contiguous Stage II Mantle Cell Lymphoma; Noncontiguous Stage II Mantle Cell Lymphoma; Stage I Mantle Cell Lymphoma; Stage III Mantle Cell Lymphoma; Stage IV Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (ibrutinib) (Experimental): Patients receive ibrutinib orally PO QD on days 1-28. Courses repeat every 28 days for up to 4 years in the absence of disease progression, unacceptable toxicity, or patient preference.
  Interventions: Drug: ibrutinib; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: ibrutinib — Given PO
  Other Names: Bruton's tyrosine kinase inhibitor PCI-32765; BTK inhibitor PCI-32765; CRA-032765; Imbruvica; PCI-32765
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This study is being done to see whether or not a drug called ibrutinib can be given to patients with mantle cell lymphoma (MCL) as maintenance therapy after induction chemotherapy. This drug blocks an enzyme that affects how the lymphocytes grow and survive. The investigators hope to learn how safe and effective ibrutinib is for treating patients with MCL after responding to induction chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the progression-free survival (PFS) rate after 3 years.

SECONDARY OBJECTIVES:

I. Assess toxicity. II. Determine rates of conversion from partial response (PR) to complete response (CR).

III. Determine median overall survival (OS) after 4 years.

TERTIARY OBJECTIVES:

I. Compare minimal residual disease (MRD) results overtime by polymerase chain reaction (PCR) and correlate these with PFS and OS.

OUTLINE:

Patients receive ibrutinib orally (PO) once daily (QD) on days 1-28. Courses repeat every 28 days for up to 4 years in the absence of disease progression, unacceptable toxicity or patient preference.

After completion of study treatment, patients who completed 4 years of treatment are followed up at 30 days. Patients who did not complete 4 years of treatment are followed up for up to 4 years post-first dose of treatment (every 3 months for 2 years and then every 6 months for 4 years).

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed mantle cell lymphoma (MCL)

  * Please note: Measurable disease is not required, but will be followed if it exists
* Patients must have received 4 or more cycles of one of the following prior systemic induction chemotherapy regimens:

  * Rituximab, cyclophosphamide, doxorubicin hydrochloride (hydroxydaunomycin), vincristine sulfate (Oncovin), prednisone (R-CHOP) (with or without alternating rituximab, dexamethasone, cytarabine [ara-c], cisplatin [platinum] [R-DHAP]) with or without autologous (auto) stem cell transplant (SCT)
  * Hyper-cyclophosphamide, vincristine sulfate, doxorubicin hydrochloride (adriamycin), dexamethasone (CVAD) with or without auto SCT
  * Bendamustine + rituximab with or without auto SCT

    * Please note:

      * Patients who received combinations of the above regimens are not eligible for enrollment
      * At the time of registration, patients must be at least 14 days out from last dose of cytotoxic chemotherapy, but no more than 90 days; if a patient underwent auto SCT, he/she must demonstrate engraftment (per treating investigator's discretion) and must meet all other hematological requirements as outlined below
* Patients must have achieved a response to induction chemotherapy (either CR or PR by Cheson 2007 criteria) and be without known progression
* Patients may have received prior radiotherapy
* Patients must exhibit an Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Absolute neutrophil count (ANC) >= 1000/mm^3, independent of growth factor support
* Platelets >= 100,000/mm^3, or >= 50,000 in cases of ongoing bone marrow involvement (in either case, these must be independent of transfusion support)
* Total bilirubin =< 1.5 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SPGT]) =< 3 x ULN
* Creatinine clearance >= 25 ml/min
* Please note: Patients who do not meet the above criteria because of Gilbert's Syndrome are still eligible
* Women of child-bearing potential (WOCBP) and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation (see timelines below for women and men); in addition, men must agree not to donate sperm during and after study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately

  * NOTE: For female patients, these restrictions apply for 1 month after the last dose of study drug; for male patients, these restrictions apply for 3 months after the last dose of study drug
  * NOTE: A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

    * Has not undergone a hysterectomy or bilateral oophorectomy; or
    * Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months)
* Female patients must have a negative pregnancy test (blood or urine) within 28 days prior to registration
* Patients must be willing and able to avoid consuming food and beverages containing grapefruit or Seville oranges while on ibrutinib study therapy
* Patients must have the ability to understand and the willingness to sign a written informed consent prior to registration on study

Exclusion Criteria:

* Patients who have received >= 7 days of prior ibrutinib or any prior treatment with another Bruton tyrosine kinase (BTK) inhibitor are not eligible
* Patients receiving ongoing treatment with any other investigational agents are not eligible
* Patients receiving live/attenuated vaccinations within 4 weeks prior to registration are not eligible
* Patients with a known central nervous system (CNS) involvement of lymphoma are not eligible (CNS staging not required)
* Patients who have undergone major surgery within 4 weeks prior to registration are not eligible
* Patients diagnosed or treated for malignancy other than MCL are not eligible unless they meet one of the following exceptions:

  * Malignancy treated with curative intent and with no known active disease present for >= 3 years before registration and felt to be at low risk for recurrence by the treating physician
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
  * Adequately treated cervical carcinoma in situ without evidence of disease
* Patients with a history of stroke or intracranial hemorrhage within 6 months prior to registration are not eligible
* Patients who require anticoagulation with warfarin or equivalent vitamin K antagonists are not eligible
* Patients who require chronic treatment with strong cytochrome P450, family 3, subfamily A, polypeptide 4/5 (CYP3A4/5) inhibitors are not eligible

  * NOTE: Patients who are currently on treatment with strong CYP3A4/5 inhibitors may be eligible if they are able to be switched to an alternative therapy that is not a strong CYP3A4/5 inhibitor prior to registration on study
* Patients with a history of allergic reactions attributed to compounds of similar chemical or biologic composition to ibrutinib are not eligible
* Patients with uncontrolled intercurrent illness including, but not limited to, any of the following are not eligible:

  * Ongoing or active systemic infection
  * Symptomatic congestive heart failure
  * Myocardial infarction within 6 months prior to registration
  * Unstable angina pectoris
  * Uncontrolled or symptomatic cardiac arrhythmias
  * Any class 3 (moderate) or class 4 (severe) cardiac disease as defined by the New York Heart Association Functional Classification
  * Psychiatric illness/social situations that would limit compliance with study requirements
* Patients who have any life-threatening illness, medical condition, or organ system dysfunction which, in the investigator's opinion, could compromise the subject's safety, interfere with the absorption or metabolism of ibrutinib capsules, or put the study outcomes at risk are not eligible
* Patients with a known human immunodeficiency virus (HIV) infection are not eligible (HIV testing not required)
* Patients with a known John Cunningham (JC) virus infection and/or progressive multifocal leukoencephalopathy (PML) are not eligible
* Patients with clinically active hepatitis A, B, or C infections are not eligible
* Female patients who are pregnant and/or lactating are not eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2015-01-12 (Actual); Primary Completion 2023-01-05 (Actual); Study Completion 2025-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Pro, MD, Principal Investigator — Northwestern University
Locations (5):
- United States (5):
  - Northwestern University, Chicago, Illinois
  - Northwestern University- Lake Forest Hospital, Lake Forest, Illinois
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Cleveland Clinic, Cleveland, Ohio
  - University of Utah, Salt Lake City, Utah

REFERENCES:
- [Derived] Karmali R, Abramson JS, Stephens DM, Barnes J, Winter JN, Ma S, Gao J, Kaplan J, Petrich AM, Hochberg E, Takvorian T, Mi X, Nelson V, Gordon LI, Pro B. Ibrutinib maintenance after frontline treatment in patients with mantle cell lymphoma. Blood Adv. 2023 Dec 12;7(23):7361-7368. doi: 10.1182/bloodadvances.2023011271. PMID 37756532

RESULTS

PARTICIPANT FLOW:
Period: Ibrutinib Treatment
Arm/Group | Treatment (Ibrutinib)
Started | 37
Cycle 1 | 36
Cycle 2 | 36
Cycle 4 | 34
Cycle 7 | 33
Cycle 13 | 30
Cycle 19 | 26
Cycle 25 | 25
Cycle 37 | 18
Cycle 49 | 17
Completed | 17
Not Completed | 20
Not completed — Adverse Event | 16
Not completed — Physician Decision | 1
Not completed — Lack of Efficacy | 1
Not completed — Death | 1
Not completed — Patient Ineligible to start treatment | 1
Period: Post Therapy Follow Up
Arm/Group | Treatment (Ibrutinib)
Started | 36
Completed | 32
Not Completed | 4
Not completed — Death | 3
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Ibrutinib)
Number analyzed (Participants) | 36
Age, Continuous [Median (Full Range); unit: years] | 60 [46 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 34
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 35
  More than one race | 0
  Unknown or Not Reported | 1
ECOG Score [Count of Participants; unit: Participants] — ECOG Performance Status
  * 0 = Fully active, able to carry on all pre-disease performance without restriction
  * 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work
  * 2 = Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  * 3 = Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours
  * 4 = Completely disabled; cannot carry on any selfcare; totally confined to bed or chair
  * 5 = Dead
  Participants
    0-1 | 34
    2 | 2
Stage at initial diagnosis [Count of Participants; unit: Participants] — Ann Arbor Staging
  * I = Localized disease, single lymph node region or single organ
  * II = Two or more lymph node regions on the same side of diaphragm
  * III = Two or more lymph node regions above and below the diaphragm
  * IV = Widespread disease; multiple organs, with or without lymph node involvement
  Participants
    I/II | 5
    III/IV | 28
    Unknown | 3
MIPI score [Count of Participants; unit: Participants] — Mantle Cell Lymphoma International Prognostic Index (MIPI) Used in patients presenting with advanced stage mantle cell lymphoma, to help prognosticate and potentially determine therapy. The score is based on 5 factors: Age, ECOG Performance Status, Serum Lactate Dehydrogenase (LDH), White Blood Cell Count, and KI-67 Proliferative Index. The total score is then classified into three categories. Low (score less than 5.7), Intermediate (Score between 5.7 and 6.2), and High (score greater than 6.2). Patients with a higher score have a poorer prognosis.
  Participants
    Low | 18
    Intermediate | 7
    High | 11
Extranodal disease at diagnosis [Count of Participants; unit: Participants] | 9
Auto-SCT consolidation prior to enrollment [Count of Participants; unit: Participants] | 18
Induction Therapy [Count of Participants; unit: Participants]
  BR | 17
  R-HyperCVAD | 9
  Nordic Regimen | 7
  R-CHOP/DHAP | 2
  R-CHOP | 1
Best response to induction therapy prior to enrollment [Count of Participants; unit: Participants]
  CR | 34
  PR | 2

OUTCOME MEASURES:

1. Primary Outcome: Determine the Progression-free Survival (PFS) Rate After 3 Years
Description: PFS will be measured from start of treatment to time of progression. Evidence of clinical progression will be documented by imaging (CT scan) for patients who have measurable disease. Progression is defined using the LUGANO Criteria, as a Deauville score of 4 or 5 (increased uptake compared to baseline) or the appearance of new lesions
Time Frame: Assessed at 3 years
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Ibrutinib)
Number analyzed (Participants) | 36
percentage of participants | 94

2. Secondary Outcome: Incidence of Adverse Events, Defined According to the National Cancer Institute's Common Terminology Criteria for Adverse Events Version 4.0
Description: To assess toxicity, all adverse events will be summarized as to type, severity, frequency, timing and attribution. Treatment related Adverse Events Occurring with Incidence of greater that or equal to 20% of patients treated with Ibrutinib Maintenance are shown here.
Time Frame: Up to 30 days after completion of study treatment, maximum 4 years post-first dose
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Ibrutinib)
Number analyzed (Participants) | 36
Participants
  Infection: Grade 1 | 4
  Infection: Grade 2 | 22
  Infection: Grade 3 | 4
  Infection: Grade 4 | 1
  Infection: Grade 0 | 5
  Lymphocyte Count Decreased: Grade 1 | 4
  Lymphocyte Count Decreased: Grade 2 | 4
  Lymphocyte Count Decreased: Grade 3 | 12
  Lymphocyte Count Decreased: Grade 4 | 9
  Lymphocyte Count Decreased: Grade 0 | 7
  White blood cells decreased: Grade 1 | 9
  White blood cells decreased: Grade 2 | 9
  White blood cells decreased: Grade 3 | 7
  White blood cells decreased: Grade 4 | 1
  White blood cells decreased: Grade 0 | 10
  Diarrhea: Grade 1 | 21
  Diarrhea: Grade 2 | 3
  Diarrhea: Grade 3 | 0
  Diarrhea: Grade 4 | 0
  Diarrhea: Grade 0 | 12
  Platelet Count Decreased: Grade 1 | 22
  Platelet Count Decreased: Grade 2 | 1
  Platelet Count Decreased: Grade 3 | 0
  Platelet Count Decreased: Grade 4 | 0
  Platelet Count Decreased: Grade 0 | 13
  Neutrophil Count Decreased: Grade 1 | 1
  Neutrophil Count Decreased: Grade 2 | 7
  Neutrophil Count Decreased: Grade 3 | 4
  Neutrophil Count Decreased: Grade 4 | 9
  Neutrophil Count Decreased: Grade 0 | 15
  Hypertension: Grade 1 | 4
  Hypertension: Grade 2 | 8
  Hypertension: Grade 3 | 8
  Hypertension: Grade 4 | 0
  Hypertension: Grade 0 | 16
  Hemorrhage: Grade 1 | 9
  Hemorrhage: Grade 2 | 4
  Hemorrhage: Grade 3 | 2
  Hemorrhage: Grade 4 | 1
  Hemorrhage: Grade 0 | 20
  Skin Rash: Grade 1 | 14
  Skin Rash: Grade 2 | 1
  Skin Rash: Grade 3 | 1
  Skin Rash: Grade 4 | 0
  Skin Rash: Grade 0 | 20
  Bruising: Grade 1 | 13
  Bruising: Grade 2 | 0
  Bruising: Grade 3 | 0
  Bruising: Grade 4 | 0
  Bruising: Grade 0 | 23
  Myalgia: Grade 1 | 10
  Myalgia: Grade 2 | 3
  Myalgia: Grade 3 | 0
  Myalgia: Grade 4 | 0
  Myalgia: Grade 0 | 23
  Fatigue: Grade 1 | 9
  Fatigue: Grade 2 | 1
  Fatigue: Grade 3 | 2
  Fatigue: Grade 4 | 0
  Fatigue: Grade 0 | 24
  Anemia: Grade 1 | 8
  Anemia: Grade 2 | 4
  Anemia: Grade 3 | 0
  Anemia: Grade 4 | 0
  Anemia: Grade 0 | 24
  Aspartate Aminotransferase increased: Grade 1 | 9
  Aspartate Aminotransferase increased: Grade 2 | 1
  Aspartate Aminotransferase increased: Grade 3 | 1
  Aspartate Aminotransferase increased: Grade 4 | 0
  Aspartate Aminotransferase increased: Grade 0 | 25
  Atrial Fibrillation/Atrial Flutter: Grade 1 | 1
  Atrial Fibrillation/Atrial Flutter: Grade 2 | 5
  Atrial Fibrillation/Atrial Flutter: Grade 3 | 4
  Atrial Fibrillation/Atrial Flutter: Grade 4 | 0
  Atrial Fibrillation/Atrial Flutter: Grade 0 | 26
  Alanine Aminotransferase increased: Grade 1 | 8
  Alanine Aminotransferase increased: Grade 2 | 0
  Alanine Aminotransferase increased: Grade 3 | 0
  Alanine Aminotransferase increased: Grade 4 | 0
  Alanine Aminotransferase increased: Grade 0 | 28

3. Secondary Outcome: Rate of Conversion From Partial Response (PR) to Complete Response (CR)
Description: Progression will be evaluated using Cheson 2007 criteria, only patients who had a PR at the time of registration and who complete ≥ 1 complete cycle of ibrutinib maintenance therapy will be evaluable for this endpoint.
Time Frame: Up to 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Ibrutinib)
Number analyzed (Participants) | 2
Participants | 1

4. Secondary Outcome: Overall Survival (OS) After 4 Years
Description: Patients will be evaluated monthly for the first 6 months on treatment, then every 3 months thereafter. Patients who go off treatment will continue to be followed for up to 4 years post-first dose. Follow-up will occur every 3 months (up to 2 years after the first dose of treatment) and then every 6 months thereafter (up to 4 years post-first dose). OS after 4 years will be calculated as a percentage of patient alive.
Time Frame: Up to 4 years post-first dose
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Ibrutinib)
Number analyzed (Participants) | 36
percentage of participants | 94

5. Other Pre Specified Outcome: Compare Minimum Residual Disease (MRD) Results Overtime by Polymerase Chain Reaction (PCR) and Correlate These With PFS and OS
Description: Archived tissue from a previous biopsy from all patients will be obtained for baseline clone identification; in addition, peripheral whole blood samples will be collected at four time points. MRD analysis will be conducted using PCR methods and results will be compared over time and correlated with PFS and OS.
Time Frame: Four time-points: baseline (pre-treatment), after 1 month and 6 months of treatment, and approximately 18-24 months post-first dose of treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: All adverse events are collected from the date of initial informed consent until 30 days after the last dose of study treatment, up to 4 years
Arm/Group | Treatment (Ibrutinib)
All-Cause Mortality (participants affected / at risk) | 4/36
Serious Adverse Events (participants affected / at risk) | 22/36
Other Adverse Events (participants affected / at risk) | 36/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Ibrutinib) (N=36)
Anemia (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 6
Atrial flutter (Cardiac disorders) | 1
Cardiac disorders - Other, specify (Cardiac disorders) | 1
Chest pain - cardiac (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 2
Ventricular fibrillation (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Rectal hemorrhage (Gastrointestinal disorders) | 1
Edema limbs (General disorders) | 1
Fatigue (General disorders) | 1
General disorders and administration site conditions - Other, specify (General disorders) | 2
Pain (General disorders) | 1
Lung infection (Infections and infestations) | 5
Pharyngitis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Skin infection (Infections and infestations) | 2
Fall (Injury, poisoning and procedural complications) | 1
Cardiac troponin I increased (Investigations) | 1
Ejection fraction decreased (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 1
White blood cell decreased (Investigations) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Transient ischemic attacks (Nervous system disorders) | 1
Confusion (Psychiatric disorders) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Social circumstances - Other, specify (Social circumstances) | 1
Hematoma (Vascular disorders) | 1
Superior vena cava syndrome (Vascular disorders) | 1
Thromboembolic event (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Ibrutinib) (N=36)
Anemia (Blood and lymphatic system disorders) | 29
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 2
Atrial flutter (Cardiac disorders) | 1
Atrioventricular block first degree (Cardiac disorders) | 1
Cardiac disorders - Other, specify (Cardiac disorders) | 4
Chest pain - cardiac (Cardiac disorders) | 3
Mobitz type I (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 4
Pericardial effusion (Cardiac disorders) | 1
Pericardial tamponade (Cardiac disorders) | 1
Sinus bradycardia (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 4
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 3
Ear pain (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Blurred vision (Eye disorders) | 1
Conjunctivitis (Eye disorders) | 1
Dry eye (Eye disorders) | 1
Eye disorders - Other, specify (Eye disorders) | 9
Keratitis (Eye disorders) | 1
Scleral disorder (Eye disorders) | 1
Vitreous hemorrhage (Eye disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 6
Anal hemorrhage (Gastrointestinal disorders) | 1
Bloating (Gastrointestinal disorders) | 2
Colitis (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 8
Diarrhea (Gastrointestinal disorders) | 27
Dry mouth (Gastrointestinal disorders) | 5
Dyspepsia (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 4
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 9
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 9
Oral hemorrhage (Gastrointestinal disorders) | 1
Oral pain (Gastrointestinal disorders) | 2
Rectal hemorrhage (Gastrointestinal disorders) | 3
Stomach pain (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 7
Chills (General disorders) | 6
Edema face (General disorders) | 2
Edema limbs (General disorders) | 12
Facial pain (General disorders) | 1
Fatigue (General disorders) | 20
Fever (General disorders) | 7
Flu like symptoms (General disorders) | 7
General disorders and administration site conditions - Other, specify (General disorders) | 9
Infusion site extravasation (General disorders) | 1
Injection site reaction (General disorders) | 1
Localized edema (General disorders) | 2
Malaise (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Pain (General disorders) | 7
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1
Allergic reaction (Immune system disorders) | 1
Autoimmune disorder (Immune system disorders) | 1
Immune system disorders - Other, specify (Immune system disorders) | 1
Bronchial infection (Infections and infestations) | 2
Eye infection (Infections and infestations) | 1
Infections and infestations - Other, specify (Infections and infestations) | 13
Laryngitis (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Otitis media (Infections and infestations) | 1
Papulopustular rash (Infections and infestations) | 1
Paronychia (Infections and infestations) | 2
Pharyngitis (Infections and infestations) | 1
Rash pustular (Infections and infestations) | 1
Rhinitis infective (Infections and infestations) | 1
Scrotal infection (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 7
Skin infection (Infections and infestations) | 3
Upper respiratory infection (Infections and infestations) | 16
Urinary tract infection (Infections and infestations) | 3
Bruising (Injury, poisoning and procedural complications) | 14
Fall (Injury, poisoning and procedural complications) | 5
Fracture (Injury, poisoning and procedural complications) | 2
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 4
Alanine aminotransferase increased (Investigations) | 13
Alkaline phosphatase increased (Investigations) | 9
Aspartate aminotransferase increased (Investigations) | 16
Blood bilirubin increased (Investigations) | 13
Cardiac troponin I increased (Investigations) | 1
Creatinine increased (Investigations) | 11
INR increased (Investigations) | 3
Investigations - Other, specify (Investigations) | 5
Lymphocyte count decreased (Investigations) | 33
Neutrophil count decreased (Investigations) | 24
Platelet count decreased (Investigations) | 28
Weight gain (Investigations) | 7
Weight loss (Investigations) | 4
White blood cell decreased (Investigations) | 29
Acidosis (Metabolism and nutrition disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 6
Dehydration (Metabolism and nutrition disorders) | 2
Glucose intolerance (Metabolism and nutrition disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 26
Hyperkalemia (Metabolism and nutrition disorders) | 7
Hypernatremia (Metabolism and nutrition disorders) | 6
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1
Hyperuricemia (Metabolism and nutrition disorders) | 5
Hypoalbuminemia (Metabolism and nutrition disorders) | 11
Hypocalcemia (Metabolism and nutrition disorders) | 14
Hypoglycemia (Metabolism and nutrition disorders) | 7
Hypokalemia (Metabolism and nutrition disorders) | 10
Hypomagnesemia (Metabolism and nutrition disorders) | 11
Hyponatremia (Metabolism and nutrition disorders) | 11
Hypophosphatemia (Metabolism and nutrition disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 6
Arthritis (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 6
Bone pain (Musculoskeletal and connective tissue disorders) | 4
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 6
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 15
Myalgia (Musculoskeletal and connective tissue disorders) | 16
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cognitive disturbance (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 10
Dysgeusia (Nervous system disorders) | 3
Headache (Nervous system disorders) | 10
Memory impairment (Nervous system disorders) | 1
Nervous system disorders - Other, specify (Nervous system disorders) | 5
Neuralgia (Nervous system disorders) | 1
Paresthesia (Nervous system disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 4
Presyncope (Nervous system disorders) | 1
Sinus pain (Nervous system disorders) | 3
Spasticity (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 3
Anxiety (Psychiatric disorders) | 2
Confusion (Psychiatric disorders) | 1
Delirium (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 3
Insomnia (Psychiatric disorders) | 3
Libido decreased (Psychiatric disorders) | 2
Psychiatric disorders - Other, specify (Psychiatric disorders) | 3
Restlessness (Psychiatric disorders) | 1
Suicidal ideation (Psychiatric disorders) | 1
Hematuria (Renal and urinary disorders) | 3
Proteinuria (Renal and urinary disorders) | 1
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1
Urinary frequency (Renal and urinary disorders) | 2
Urinary retention (Renal and urinary disorders) | 1
Urinary urgency (Renal and urinary disorders) | 2
Pelvic pain (Reproductive system and breast disorders) | 3
Prostatic obstruction (Reproductive system and breast disorders) | 2
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 2
Vaginal hemorrhage (Reproductive system and breast disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 17
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 13
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 11
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 8
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 5
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2
Nail discoloration (Skin and subcutaneous tissue disorders) | 1
Nail ridging (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Purpura (Skin and subcutaneous tissue disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 12
Scalp pain (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 18
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 1
Flushing (Vascular disorders) | 1
Hematoma (Vascular disorders) | 4
Hot flashes (Vascular disorders) | 2
Hypertension (Vascular disorders) | 27
Hypotension (Vascular disorders) | 2
Superior vena cava syndrome (Vascular disorders) | 1
Thromboembolic event (Vascular disorders) | 3
Vascular disorders - Other, specify (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-03): https://cdn.clinicaltrials.gov/large-docs/97/NCT02242097/Prot_SAP_000.pdf